CLINICAL TRIAL: NCT03117946
Title: Modulation of Anti-tumor T Cell Responses in Cancer Patients Treated by Concomitant Radiochemotherapy
Acronym: i-RTCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: API/2016/67
Record Dates: First submitted 2017-04-13; First posted 2017-04-18 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Lung Cancer; Head and Neck Cancer
Keywords: immunomonitoring; immune checkpoint; chemoradiation; T cells
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Biological samples (Experimental): Blood samples will be collected at baseline, at J15/J20 after RTCT initiation, and then 1 month, 3 months and 12 months after the end of RTCT treatment, and at disease progression if applicable.
  Tumor tissues will be collected if available.
  Interventions: Other: Biological samples

INTERVENTIONS:
Other: Biological samples — blood and tumor tissue sample

SUMMARY:
The aim of this study is to evaluate modulation of anti-tumor T cell responses in cancer patients treated by concomitant radiochemotherapy (i-RTCT)

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed NSCLC (Non Small Cell Lung Cancer) or SCLC (small cell lung cancer) OR histologically confirmed Head and neck cancer
* Patient candidate to a first-line concomitant radiochemotherapy
* Written informed consent

Exclusion Criteria:

* Sequential radiochemotherapy, exclusive radiotherapy, or stereotactic radiotherapy
* History of adjuvant radiochemotherapy for cancer treatment
* Patients under immunotherapy, chemotherapy or other immunosuppressive drugs (prednisone or prednisolone ≤ 10 mg/day is allowed)
* HIV, hepatitis C or B virus
* Patients with any medical or psychiatric condition or disease,
* Patients under guardianship, curatorship or under the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2017-05-29 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-11-29 (Estimated)

PRIMARY OUTCOMES:
tumor antigen specific T-cell responses | up to 12 months after the end of radiochemotherapy
  tumor antigen specific T-cell responses

SECONDARY OUTCOMES:
monitoring of immune checkpoints, immune cell death, immune suppressive cells and T-cell polarisation | up to 12 months after the end of radiochemotherapy
  monitoring of immune checkpoints, immune cell death, immune suppressive cells and T-cell polarisation
Progression free survival | date of first progression of the disease (within 2 year after the initiation of the treatment)]
  time interval between the date of initiation of treatment and the date of first progression (local, remote [extent of the disease by RECIST v1.1] second cancer) or death from any cause
overall survival | date of death from any cause (within 2 years after the initiation of the treatment)
  time between the date of initiation of treatment and the date of death from any cause
Quality of life related to health measured by EORTC-QLQC30 | from the inclusion to patient death, up to 1 year
  Quality of life related to health measured by EORTC-QLQC30

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Besançon, Besançon
  - Centre Georges François LECLERC, Dijon
  - Hôpital Nord Franche-Comté, Montbéliard
  - Institut Jean Godinot, Reims